CLINICAL TRIAL: NCT00551122
Title: Phase I/II Multicentre Trial of Salvage Chemotherapy With Gem-TIP for Relapsed Germ Cell Cancer
Brief Title: Gemcitabine, Paclitaxel, Ifosfamide, and Cisplatin in Treating Patients With Progressive or Relapsed Metastatic Germ Cell Tumors
Acronym: GemTIP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000572096; USCTU-UR1002-GEM-TIP; EU-20769; EUDRACT-2004-004804-19
Record Dates: First submitted 2007-10-25; First posted 2007-10-30 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2007-10

CONDITIONS: Brain and Central Nervous System Tumors; Extragonadal Germ Cell Tumor; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; testicular seminoma; recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; stage III malignant testicular germ cell tumor; testicular choriocarcinoma and seminoma; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular yolk sac tumor and teratoma with seminoma; recurrent extragonadal non-seminomatous germ cell tumor; recurrent extragonadal seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; recurrent extragonadal germ cell tumor; ovarian mixed germ cell tumor; adult central nervous system germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma; Endodermal Sinus Tumor | interventions — Filgrastim; Lenograstim; pegfilgrastim; Cisplatin; Gemcitabine; Ifosfamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel, gemcitabine, cisplatin, ifosfamide (Experimental): Day 1 Dexamethasone sodium phosphate 25mg I/V ) before Chlorphenamine 10mg I/V 30 - 60 mins ) paclitaxel Ranitidine 50mg I/V ) Paclitaxel - 175 mg m2 I/V in 500ml normal saline over 3 hours Gemcitabine - 1200mg per m2 I/V in 500ml normal saline over 30 mins Days 1-5 Cisplatin 20mg per m2 in 1 litre normal saline over 4 hours 2 litres normal saline over 16 hours, each litre containing 10 mmol MgSO4 and 20mmol KCL.
  If urine output is insufficient (less than 600ml per 6 hours) or if excessive weight gain (greater than 2kg) 100 - 200ml 10% mannitol should be used. Alternatively, low dose frusemide (20mg I/V) can be used.
  Days 2 - 6 Ifosfamide 1G per m2 + MESNA 0.5G m2 in 500 ml normal saline over 1 hour after the cisplatin infusion.
  MESNA 0.5G m2 to be included in first 1 litre post cisplatin hydration bag Pegylated G-CSF will be given on day 7 as an alternative to daily G-CSF.
  Interventions: Biological: filgrastim; Biological: lenograstim; Biological: pegfilgrastim; Drug: cisplatin; Drug: gemcitabine hydrochloride; Drug: ifosfamide; Drug: paclitaxel

INTERVENTIONS:
Biological: filgrastim
Biological: lenograstim
Biological: pegfilgrastim
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: ifosfamide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, paclitaxel, ifosfamide, and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of gemcitabine when given together with paclitaxel, ifosfamide, and cisplatin, and to see how well they work in treating patients with progressive or relapsed metastatic germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose (MTD) of gemcitabine hydrochloride when administered with TIP chemotherapy comprising paclitaxel, ifosfamide, and cisplatin with growth factor support (Gem-TIP) in patients with progressive or relapsed metastatic germ cell tumors.
* To compare the MTD of the Gem-TIP regimen with the MTD determined in a previous Medical Research Council study of TIP alone.
* To compare the degree of dose intensification achieved with Gem-TIP chemotherapy with that achieved in the prior study of TIP chemotherapy alone.
* To assess the dose of gemcitabine hydrochloride that can be delivered with the TIP regimen in these patients.
* To measure response rates and failure-free survival of patients treated with Gem-TIP alone.
* To assess the utility of PET scanning after Gem-TIP chemotherapy in these patients.

OUTLINE: This is a multicenter, phase I dose-escalation study of gemcitabine hydrochloride followed by a phase II study.

* Phase I: Patients receive gemcitabine hydrochloride IV over 30 minutes and paclitaxel IV over 3 hours on day 1, cisplatin IV over 4 hours on days 1-5, and ifosfamide IV over 1 hour on days 2-6. Patients also receive filgrastim or lenograstim (G-CSF) subcutaneously (SC) on days 7-18 or until blood counts recover OR pegfilgrastim SC once on day 6. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Phase II: An additional cohort of 14 patients is treated as in phase I at the MTD determined in phase I.

After completion of study therapy, patients are followed periodically for up to 1 year and then at the investigator's discretion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets the following criteria:

  * Histologically confirmed extracranial primary germ cell cancer, seminoma, or nonseminoma

    * Unresectable metastatic disease
    * No completely resected cancer
  * Rising serum markers (i.e., alpha-fetoprotein and human chorionic gonadotropin) on sequential measurement or biopsy-proven unresectable germ cell cancer
* In first relapse after a single prior cisplatin-containing combination chemotherapy

  * Patients with late relapse (i.e., > 2 years post initial chemotherapy) should be considered for surgery rather than chemotherapy, if technically feasible
* No patients with cerebral metastases alone

  * Progressive cerebral and systemic disease may be considered for this study, provided cranial irradiation is also considered as a component of care

PATIENT CHARACTERISTICS:

* Medically and psychologically fit to receive this intensive chemotherapy schedule
* WBC > 3.5 times 10^9/L
* Platelet count > 130 times 10^9/L
* Glomerular filtration rate ≥ 50 mL/min (as determined by 24 hour creatinine clearance or nuclear medicine technique)
* Fertile patients must use effective contraception
* No other prior malignancy except successfully treated nonmelanoma skin cancer or superficial bladder cancer
* No prior allergic reactions to cisplatin or other platinum compounds

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2006-11; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of gemcitabine hydrochloride when administered with TIP chemotherapy comprising paclitaxel, ifosfamide, and cisplatin with growth factor support (phase I) | end of study
Response rates (phase I) | end of study
Failure-free survival (phase I) | end of study
Utility of positron emission tomography scanning after Gem-TIP chemotherapy (phase I) | end of study
Degree of dose intensification achieved with Gem-TIP chemotherapy relative to a previous Medical Research Council study with TIP alone (phase II) | end of study

CONTACTS AND LOCATIONS:
Overall Officials: G. Mead, MD, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England